CLINICAL TRIAL: NCT06824610
Title: The Effect of Different Oxygen Flow Rates on End-tidal Carbon Dioxide Monitoring During Procedural Sedation in Patients Undergoing Minor Gynaecological Procedures.
Brief Title: The Effect of Oxygen Flow Rate on End-tidal CO2 During Deep Sedation
Status: Not yet recruiting | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Marina Adel Karam Lemoun, Principal Investigator Marina A. K. Lemoun, Minia University
Other Study IDs: use of capnography in sedation
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Capnography
MeSH Terms: interventions — Capnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group A: received 4 L /min oxygen flow rate.
  Interventions: Device: capnography
- Group B: received 6 L /min oxygen flow rate.
  Interventions: Device: capnography
- Group C: received 8 L /min oxygen flow rate.
  Interventions: Device: capnography

INTERVENTIONS:
Device: capnography — measurment of end-tidal carbon dioxide

SUMMARY:
This study aims to detect the effect of different O2 flow rates on end tidal carbon dioxide level in patients scheduled for minor gynaecological procedures under deep sedation using laryngeal mask airway.

* Primary outcome was measuring end tidal carbon dioxide ( EtCO2 ) non invasively by laryngeal mask all through the procedure.
* Secondary outcomes included peripheral O2 saturation, hemodynamics, time to recovery, total propofol dose, patients' satisfaction, sedation score, and complications.

DETAILED DESCRIPTION:
Procedural sedation (PS) is generally considered to include the stages of moderate and deep sedation of the continuum of anaesthesia . The clinical goals of procedural sedation are to alleviate apprehension, ameliorate the examination, findings, minimize the patients' memories of the incident and to control pain and distress during diagnostic and interventional medical procedures a lot of minor gynaecological procedures can be performed under moderate to deep sedation as ( D&C Biopsy, hysteroscopic polypectomy and diagnostic hysteroscopies ) The greatest threat to the safety of sedated patient is airway compromise and or respiratory depression . To decrease the risk of airway and respiratory complications, careful attention must be directed toward the appropriate selection of medications, adherence to dosing recommendations, and most importantly the identification of the high-risk patient.

Regardless of the clinical scenario or the medications used, appropriate monitoring of the patient's respiratory and physiologic functions is mandatory to rapidly identify respiratory compromise.

Respiratory function is usually evaluated by observation of qualitative clinical signs (respiratory rate, depth and effort) and oxygen saturation monitoring. Oxygen desaturation in pulse oximetry usually occurs as a delayed sign , so if the capnograph monitor is used, any increase in EtCO2 during hypoventilation can alert the observing anesthetist to avoid hypoxemia. Capnography is a respiratory monitoring device that has become an accepted standard of care for PS in many circumstances. So, the American Society of Anesthesiology standards for Basic Anesthetic Monitoring require the use of capnography for both moderate and deep sedation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 18-45 years
2. ASA physical status l : ll
3. Minor elective gynaecological procedures lasting less than 30 minutes ( D&C biopsy, hysteroscopic polypectomy and diagnostic hysteroscopy )

Exclusion Criteria:

* We will exclude from the study patients with the following:

  1. Patient refusal to participate in this study.
  2. ASA lll or more.
  3. Lengthy procedures taking more than 30 minutes
  4. Contraindication for the use of laryngeal mask airway as ( pharyngeal pathology, risk of aspiration and airway obstruction below larynx)
  5. BMI more than 35

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: females aged between18 - 45 years old scheduled for minor gynaecological procedures under deep sedation
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
carbon dioxide monitoring | baseline and every 5 minutes all through the procedure
  Primary outcome is measuring end tidal carbon dioxide ( EtCO2 ) non invasively by laryngeal mask all through the procedure.

SECONDARY OUTCOMES:
peripheral O2 saturation | baseline and every 5 minutes all through the procedure
  peripheral O2 saturation

CONTACTS AND LOCATIONS:
Overall Officials: Marina A Karam Lemoun, Master, Principal Investigator — Minia University

IPD SHARING:
Plan to Share IPD: No
Data is available with a corresponding author on reasonable request

REFERENCES:
- [Background] Askar H, Misch J, Chen Z, Chadha S, Wang HL. Capnography monitoring in procedural intravenous sedation: a systematic review and meta-analysis. Clin Oral Investig. 2020 Nov;24(11):3761-3770. doi: 10.1007/s00784-020-03395-1. Epub 2020 Jun 16. PMID 32556657
- [Background] Wadhwa V, Gupta K, Vargo JJ. Monitoring standards in sedation and analgesia: the odyssey of capnography in sedation for gastroenterology procedures. Curr Opin Anaesthesiol. 2019 Aug;32(4):453-456. doi: 10.1097/ACO.0000000000000756. PMID 31169549
- [Background] Dewdney C, MacDougall M, Blackburn R, Lloyd G, Gray A. Capnography for procedural sedation in the ED: a systematic review. Emerg Med J. 2017 Jul;34(7):476-484. doi: 10.1136/emermed-2015-204944. Epub 2016 Aug 26. PMID 27565194